CLINICAL TRIAL: NCT00095823
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Aripiprazole as Adjunctive Therapy in the Treatment of Patients With Major Depressive Disorder.
Brief Title: A Study of Adjunctive Aripiprazole in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-139
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Antidepressive Agents; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- A1 (Placebo Comparator)
  Interventions: Drug: Antidepressant + Placebo
- A2 (Active Comparator)
  Interventions: Drug: Antidepressant + Aripiprazole
- A3 (No Intervention)

INTERVENTIONS:
Drug: Antidepressant + Placebo — Antidepressant Caps/Tablets Placebo Tablets, Oral, 2-20 mg Placebo, once daily, 6 weeks following an 8 week Prospective Treatment (Baseline) Phase.
  Arms: A1
Drug: Antidepressant + Aripiprazole — Antidepressant Caps/Tablets Aripiprazole Tablets, Oral, 2-20 mg Aripiprazole, once daily, 6 weeks following an 8 week Prospective Treatment (Baseline) Phase.
  Other Names: Abilify
  Arms: A2

SUMMARY:
This trial is a 14 week, randomized, double-blind, placebo controlled study, to assess the safety and efficacy of aripiprazole as adjunctive treatment to an ongoing antidepressant treatment in patients with Major Depressive Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-65 years old
* Experienced a Major Depressive Disorder with the current episode of minimally 8 weeks in duration.
* Treatment history of an inadequate response to at least one and no more than three antidepressants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 2004-06; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Change in a depression rating scale at endpoint

SECONDARY OUTCOMES:
Change in a disability scale and Clinical Global Impression scale at endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- United States (20):
  - Local Institution, Garden Grove, California
  - Local Institution, Northridge, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Jacksonville, Florida
  - Local Institution, Chicago, Illinois
  - Local Institution, Edwardsville, Illinois
  - Local Institution, Rockville, Maryland
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Farmington Hills, Michigan
  - Local Institution, Okemos, Michigan
  - Local Institution, Staten Island, New York
  - Local Institution, Portland, Oregon
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Austin, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Woodstock, Vermont
  - Local Institution, Charlottesville, Virginia
  - Local Institution, Bellevue, Washington
  - Local Institution, Seattle, Washington
  - Local Institution, Middleton, Wisconsin

REFERENCES:
- [Derived] Stewart TD, Hatch A, Largay K, Sheehan JJ, Marler SV, Berman RM, Nelson JC. Effect of symptom severity on efficacy and safety of aripiprazole adjunctive to antidepressant monotherapy in major depressive disorder: a pooled analysis. J Affect Disord. 2014 Jun;162:20-5. doi: 10.1016/j.jad.2014.03.017. Epub 2014 Mar 24. PMID 24766999
- [Derived] Fabian TJ, Cain ZJ, Ammerman D, Eudicone JM, Tang Y, Rollin LM, Forbes RA, Berman RM, Baker RA. Improvement in functional outcomes with adjunctive aripiprazole versus placebo in major depressive disorder: a pooled post hoc analysis of 3 short-term studies. Prim Care Companion CNS Disord. 2012;14(6):PCC.12m01394. doi: 10.4088/PCC.12m01394. Epub 2012 Dec 20. PMID 23585999
- [Derived] Dunner DL, Laubmeier KK, Manos G, Forbes RA, Baker RA, Berman RM. Beneficial effects of adjunctive aripiprazole in major depressive disorder are not dependent on antidepressant therapy history: a post hoc analysis of 3 randomized, double-blind, placebo-controlled trials. Prim Care Companion CNS Disord. 2012;14(6):PCC.12m01380. doi: 10.4088/PCC.12m01380. Epub 2012 Nov 22. PMID 23585997
- [Derived] Casey DE, Laubmeier KK, Marler SV, Forbes RA, Baker RA. Efficacy of adjunctive aripiprazole in major depressive disorder: a pooled response quartile analysis and the predictive value of week 2 early response. Prim Care Companion CNS Disord. 2012;14(3):PCC.11m01251. doi: 10.4088/PCC.11m01251. Epub 2012 May 31. PMID 23106023
- [Derived] Fava M, Dording CM, Baker RA, Mankoski R, Tran QV, Forbes RA, Eudicone JM, Owen R, Berman RM. Effects of adjunctive aripiprazole on sexual functioning in patients with major depressive disorder and an inadequate response to standard antidepressant monotherapy: a post hoc analysis of 3 randomized, double-blind, placebo-controlled studies. Prim Care Companion CNS Disord. 2011;13(1):PCC.10m00994. doi: 10.4088/PCC.10m00994gre. PMID 21731833
- [Derived] Weisler RH, Khan A, Trivedi MH, Yang H, Eudicone JM, Pikalov A, Tran QV, Berman RM, Carlson BX. Analysis of suicidality in pooled data from 2 double-blind, placebo-controlled aripiprazole adjunctive therapy trials in major depressive disorder. J Clin Psychiatry. 2011 Apr;72(4):548-55. doi: 10.4088/JCP.09m05495gre. Epub 2010 Aug 24. PMID 20816039
- [Derived] Nelson JC, Thase ME, Trivedi MH, Fava M, Han J, Van Tran Q, Pikalov A, Qi Y, Carlson BX, Marcus RN, Berman RM. Safety and Tolerability of Adjunctive Aripiprazole in Major Depressive Disorder: A Pooled Post Hoc Analysis (studies CN138-139 and CN138-163). Prim Care Companion J Clin Psychiatry. 2009;11(6):344-52. doi: 10.4088/PCC.08m00744gre. PMID 20098527
- [Derived] Thase ME, Trivedi MH, Nelson JC, Fava M, Swanink R, Tran QV, Pikalov A, Yang H, Carlson BX, Marcus RN, Berman RM. Examining the efficacy of adjunctive aripiprazole in major depressive disorder: a pooled analysis of 2 studies. Prim Care Companion J Clin Psychiatry. 2008;10(6):440-7. doi: 10.4088/pcc.v10n0603. PMID 19287552
- [Derived] Trivedi MH, Thase ME, Fava M, Nelson CJ, Yang H, Qi Y, Tran QV, Pikalov A, Carlson BX, Marcus RN, Berman RM. Adjunctive aripiprazole in major depressive disorder: analysis of efficacy and safety in patients with anxious and atypical features. J Clin Psychiatry. 2008 Dec;69(12):1928-36. Epub 2008 Dec 2. PMID 19192475
- [Derived] Boulton DW, Balch AH, Royzman K, Patel CG, Berman RM, Mallikaarjun S, Reeves RA. The pharmacokinetics of standard antidepressants with aripiprazole as adjunctive therapy: studies in healthy subjects and in patients with major depressive disorder. J Psychopharmacol. 2010 Apr;24(4):537-46. doi: 10.1177/0269881108096522. Epub 2008 Oct 2. PMID 18832427
- [Derived] Berman RM, Marcus RN, Swanink R, McQuade RD, Carson WH, Corey-Lisle PK, Khan A. The efficacy and safety of aripiprazole as adjunctive therapy in major depressive disorder: a multicenter, randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2007 Jun;68(6):843-53. doi: 10.4088/jcp.v68n0604. PMID 17592907